CLINICAL TRIAL: NCT07223346
Title: Latinas Integrating Fitness and Therapy (LIFT)
Brief Title: Latinas Integrating Fitness and Therapy
Acronym: LIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Jessica Gonzalez, Associate Professor, Colorado State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 6710; Pilot Grant (Other: University of Colorado Cancer Center)
Record Dates: First submitted 2025-07-25; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Stepped Care Cognitive Behavioral Therapy; Exercise; Physical Activity; Anxiety Depression
Keywords: Latina cancer survivors; Mental health counseling; Stepped-care; Exercise; Physical activity
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combining exercise program and stepped-care counseling (Experimental): Investigators are offering Latinas who have cancer a combination of an exercise program and mental health that will take place online. All participants will receive an 8 week evidence-based exercise program. In addition, Latinas with cancer will take a survey on depression and anxiety to determine which level of mental counseling they will receive. They will take surveys at 2 weeks, 6 weeks, and 10 weeks to see if their levels of depression and anxiety have changed. If their symptoms increase they will receive more counseling sessions.
  Interventions: Behavioral: Stepped Care Mental Health Counseling; Behavioral: Exercise Program

INTERVENTIONS:
Behavioral: Stepped Care Mental Health Counseling — Counseling Sessions: Everyone will have one orientation session with a counselor to learn about the study. After that, based on their levels of anxiety and depression, they may get between 1 and 7 counseling sessions. Milder levels of depression and anxiety will receive fewer sessions. The counseling sessions can include a self-help guide, coping strategies, self-help tips, and a type of therapy called cognitive behavioral therapy (CBT), which is specially adapted for Latina cancer survivors. The counseling sessions will take place online via zoom.
  Other Names: AYUDA
Behavioral: Exercise Program — The exercise program consists of easy to moderate aerobic and resistance training and discussions about staying active. These sessions will take place in your home, on zoom, led by a qualified exercise professional, and may be held in a group with other Latina cancer survivors. They will receive exercise equipment to use during the study and keep after the study ends. Exercise sessions are once per week for about an hour, and the discussion sessions take place before or after three of these sessions, and last about 30-45 minutes. If they miss a session or want to review, they will have access to recorded videos.
  Other Names: FitCancer

SUMMARY:
Investigators are studying how combining a stepped-care mental health counseling program with an evidence-based exercise program can help Latina cancer survivors feel better mentally and physically. The goal is to improve stress, emotions, and physical activity during and after cancer treatment. In addition, investigators will examine the feasibility and acceptability of the intervention among Latina cancer survivors.

DETAILED DESCRIPTION:
This study will be 10 weeks and offered online via Zoom. Participants can choose for their exercise and counseling sessions and materials to be in English or Spanish. If participants join they will: (1) Complete surveys at the beginning, 2 weeks, 6 weeks, and 10 weeks. These may consist of questions asking about levels of anxiety and depression, physical activity, and quality of life. (2) At week 1 and week 10, be asked to complete assessments of physical ability, which include muscular endurance and balance. (3) Participate in an 8-week evidence-based exercise program, which includes: one-hour exercise session 1 time per week and three, 30-minute discussion sessions to help them stay active after the study ends. (4) Receive one orientation meeting the counselor and up to seven one-hour individual counseling sessions with a counselor who will be supervised by a licensed therapist. The number of counseling sessions received will depend on their feelings or symptoms of anxiety or depression. If these symptoms are mild, they will receive fewer sessions. Counseling session will last approximately 1-hour and be online. (5) Counseling, exercise, and discussion sessions will be recorded for training purposes, but will keep identities private. (6) The total time commitment will be between 1-3 hours per week, for 8-weeks.

ELIGIBILITY:
Inclusion Criteria: 1) currently undergoing or within 6-months of completing primary cancer(s) (2) self-identify as Latina and female, (3) over the age of 18 years, (4) reside in Colorado, (4) have access to internet, and be (5) English or Spanish speaking.

Exclusion Criteria: (1) metastatic disease, (2) known contraindications for exercise (e.g. existing CVD or metabolic disease, use of an assistive-walking device, severe ataxia, etc.), (3) part of a vulnerable population (pregnant, homeless, in prison, have auditory impairment), and (4) currently participating in mental health counseling with a licensed professional and/or a structured exercise program.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of LIFT intervention components | At the completion of the study of the individual's exercise and counseling program.
  Feasibility will include the rate of recruitment, participant retention, and completeness of data. Acceptability, among participants (i.e., cancer survivors) will be assessed via survey and focus groups.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) | Administered at baseline, week 2, 6, and 10.
  The PROMIS short forms for depression and anxiety are used to measure how often a person has felt symptoms such as sadness, worry, or nervousness during the past 7 days. Each form includes 8 questions with answers ranging from 1 ("Never") to 5 ("Always"). Scores can range from 8 to 40, with higher scores meaning more depression or anxiety symptoms.
Functional Assessment of Cancer Therapy -General (FACT-G) | Administered at baseline and week 10.
  The FACT-G is a 27-item questionnaire used to assess health-related quality of life in people with cancer. It includes four subscales: Physical Well-Being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB), and Functional Well-Being (FWB). Scores for each subscale are calculated by adding the responses, with adjustments made for any missing items. These subscale scores are then combined to produce a total FACT-G score. The total score ranges from 0 to 108, with PWB, SWB, and FWB each ranging from 0-28, and EWB ranging from 0-24. Higher scores indicate a better quality of life.
Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Administered at baseline and week 10.
  Description: The GLTEQ is a self-reported questionnaire used to assess the frequency and duration of aerobic and strength-based physical activity during leisure time over the past month. Participants report how many days per week and how many minutes per session they engage in light, moderate, and vigorous aerobic exercise, as well as strength or resistance training. Only sessions lasting 10 minutes or more and performed during free time are included. The questionnaire also asks about the average time spent sitting on weekdays. Moderate-to-vigorous physical activity (MVPA) and moderate-to-vigorous physical activity including resistance and aerobic activities (MVPA R+A) are calculated by combining the frequency and duration of moderate and vigorous sessions. Higher values indicate greater physical activity.
International Physical Activity Questionnaire (IPAQ) | Administered at baseline and week 10.
  The IPAQ Short Form is a self-reported questionnaire that assesses physical activity levels over the previous 7 days. It asks about the frequency and duration of vigorous activity, moderate activity, walking, and sedentary behavior. Participants report the number of days they engaged in each activity for at least 10 minutes at a time, along with the hours and minutes spent on those days. These responses can be combined into a total number of minutes per week to represent overall physical activity (for example, 3 hours equal to 180 minutes) or reported as hours and minutes (for example, 2 hours and 20 minutes). Sedentary behavior is measured separately by asking about total sitting or lying down time on a typical weekday, also recorded in hours and minutes. Scores range from 0 minutes per week with no maximum limit, and higher scores indicate greater physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Gonzalez-Voller, Ph.D, Principal Investigator — Colorado State University; Heather Leach, Ph.D, Principal Investigator — Colorado State University
Locations (1):
- Colorado State Univerisity, Fort Collins, Colorado, United States

REFERENCES:
- [Background] Leach HJ, Mama SK, Harden SM. Group-based exercise interventions for increasing physical activity in cancer survivors: a systematic review of face-to-face randomized and non-randomized trials. Support Care Cancer. 2019 May;27(5):1601-1612. doi: 10.1007/s00520-019-04670-y. Epub 2019 Feb 9. PMID 30739169
- [Background] Leach HJ, Crisafio ME, Howell MJ, Nicklawsky A, Marker RJ. A Group-Based, Videoconference-Delivered Physical Activity Program for Cancer Survivors. Transl J Am Coll Sports Med. 2023 Spring;8(2):e000221. doi: 10.1249/tjx.0000000000000221. Epub 2023 Feb 10. PMID 37974897
- [Background] Gonzalez-Voller, J., Schumacher, A. R., Nguyen, J., Kilbourn, K., Okuyama, S., Fullwood, C. R., & Borrayo, E. A. (2025). The AYUDA Pilot-Study Intervention: Psychosocial Support for Underserved Spanish-Speaking Latinas Undergoing Breast Cancer Treatment. Hispanic Journal of Behavioral Sciences, 0(0). https://doi.org/10.1177/07399863251357733